CLINICAL TRIAL: NCT00195468
Title: A Randomized, Open-label Study to Compare the Safety and Efficacy of Cyclosporine Dose Reduction With Cyclosporine Elimination in De Novo Renal Allograft Recipients Receiving Rapamune.
Brief Title: Study Comparing Cyclosporine Dose Reduction vs. Cyclosporine Elimination in Kidney Transplant Recipients Taking Sirolimus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468H1-101116
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2007-12

CONDITIONS: Kidney Failure; Graft vs Host Disease
Keywords: Kidney Failure; Transplant
MeSH Terms: conditions — Renal Insufficiency; Graft vs Host Disease | interventions — Cyclosporine

INTERVENTIONS:
Drug: CYCLOSPORINE

SUMMARY:
Compare kidney function as measured by calculated creatinine clearance (using the method by Nankivell)1 at 12 months after transplantation in subjects receiving induction therapy with cyclosporine microemulsion (CsA) and Rapamune followed by CsA dose reduction (Group I) with subjects receiving induction therapy with CsA and Rapamune followed by CsA discontinuation (Group II).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with end-stage renal disease scheduled to receive a primary or secondary renal allograft from a cadaveric donor, from a living-unrelated donor, or a living-related HLA-mismatched donor. Subjects must be at least 18 years of age.

Exclusion Criteria:

* Subjects with active major infection, including active hepatitis B or C infection, decreased platelets, elevated lipids, or multiple organ transplants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2004-03; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Calculated creatinine clearance at 12 months post transplantation for patients on therapy.

SECONDARY OUTCOMES:
Calculated creatinine clearance at 6 months Serum creatinine at 6 and 12 months post-transplantation. Graft survival at 6 and 12 months post-transplantation. Incidence of biopsy confirmed acute graft rejections at 6 and 12 months post transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Brazil, xavierl@wyeth.com; Trial Manager, Principal Investigator — For Mexico, gomezlj@wyeth.com
Locations (9):
- Brazil (6):
  - Curitiba, Paraná
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Ribeirao Preto, Rio Grande do Sul
  - São José do Rio Preto, São Paulo
  - São Paulo, São Paulo
- Mexico (3):
  - Chihuahua City, Chihuahua
  - Torreón, Coahuila
  - Mexico City DF